CLINICAL TRIAL: NCT05102487
Title: Patient Comprehension, Retention and Satisfaction With Anesthesia Consent Process
Brief Title: Anesthesia Consent Process
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated early
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB21-1573
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia Risks; Anesthesia Consent; Anesthesia; Consent Retention; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently at University of Chicago Medical Center (UCMC) consent for anesthesia is obtained verbally by qualified anesthesia providers. Later this year, the investigators will be moving to a written informed consent form for anesthesia that must be signed by patients before proceeding with elective surgery. The department's aim is to study patient satisfaction and retention of information presented before and after this change is made.

After consent for anesthesia is obtained, study personnel will approach patients >= 18 years of age scheduled for elective surgery and, after seeking verbal consent for this study, will administer a questionnaire which will assess patient satisfaction and retention of the risks that were presented.

DETAILED DESCRIPTION:
Currently at UCMC consent for anesthesia is obtained verbally by qualified anesthesia providers. Later this year, the investigators will be moving to a written informed consent form for anesthesia that must be signed by patients before proceeded with elective surgery. The aim is to study patient satisfaction and retention of information presented before and after this change is made.

Study Procedures After consent for anesthesia is obtained, study personnel will approach patients >= 18 years of age scheduled for elective surgery and, after seeking verbal consent for this study, will administer a questionnaire which will assess patient satisfaction and retention of the risks that were presented.

Demographic data will be recorded, including age, sex, classification of surgery (by service), urgency of case, as well as role of person obtaining anesthesia consent (resident vs. CRNA/APN vs. attending anesthesiologist). Method of obtaining anesthesia consent will also be recorded. Patient identifiers, including name, MRN and date of birth will NOT be recorded as part of this study.

Patients will be approached for participation in this study preoperatively, in the pre-op holding area, immediately after anesthesia consent is obtained by the appropriate anesthesia provider. The patient's electronic medical record will NOT be accessed in order to pre-screen for participation no PHI will be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking Age> 18 years old

Exclusion Criteria:

* Emergency cases Pt unable to consent for themselves Age <18 yo Pregnant women for delivery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All anesthesia cases that fit the criteria above will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Upon receiving consent for anesthesia, pre-operatively
  How well patients are satisfied with the anesthesia consent process by using a 6 question questionnaire developed for this study.

SECONDARY OUTCOMES:
Patient Retention | Upon receiving consent for anesthesia, pre-operatively
  How well the patient was able to retain the information disclosed during the anesthesia by consent by using a 6 question questionnaire developed for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Junaid Nizamuddin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States